CLINICAL TRIAL: NCT05403970
Title: Correlation of Various Laboratory Parameters With Outcome in Patients Suffering From Acute Non-traumatic Subarachnoid Hemorrhage - Prospective Case Series
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Tamas Vegh, MD, associate professor, University of Debrecen
Other Study IDs: DE KK RKEB/IKEB 5924-2021
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Subarachnoid Hemorrhage
Keywords: subarachnoid hemorrhage; anemia; vasospasm; vitamin D; modified clot lysis assay
MeSH Terms: conditions — Subarachnoid Hemorrhage; Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective study, the investigators aim to investigate the effect of the following three factors on the development of vasospasm and patient outcome: (1.) the role of anemia; (2.) the role of plasma fibrinolytic activity; (3.) the role of vitamin D.

The investigators include patients admitted to the Neurosurgical Intensive Care Unit of the Clinical Center of the University of Debrecen with the diagnosis of subarachnoid hemorrhage (SAH). Patients are treated according to international guidelines. As part of the study protocol the following investigations are performed: • Hemoglobin level measurement: on the day of admission and day 3-4-7 and 14 after hemorrhage •Modified clot lysis assay (mCLA): on the day of admission and day 7 after hemorrhage •25-hydroxy vitamin-D level measurement: on the day of admission •Transcranial color-coded duplex sonography (detecting vasospasm): on daily basis. •30 day follow-up: mortality, Glasgow Outcome Scale (GOS), Karnofsky score, Barthel score •90 day follow-up: mortality, Glasgow Outcome Scale , Karnofsky score, Barthel score. Laboratory test results are correlated with (a) the development of vasospasm; (b) with 30 and 90 day outcome.

Perspectives of the planned study: Considering the currently available therapeutic range for patients with SAH, results of the present study may provide a basis for designing further randomized, prospective trials to investigate the effect of treating anemia, anticoagulation and vitamin-D supplementation.

DETAILED DESCRIPTION:
Background

The incidence of aneurysmal subarachnoid hemorrhage is 10/100000 person/year. Some epidemiological date suggest that the 30-day mortality of subarachnoid hemorrhage (SAH) is nearly 50%. (ACROSS Group. Epidemiology of aneurysmal subarachnoid hemorrhage in Australia and New Zealand: incidence and case fatality from the Australasian Cooperative Research on Sub- arachnoid Hemorrhage Study (ACROSS). Stroke. 2000;31: 1843-50 Ingall T, Asplund K, Mahonen M, Bonita R. A multinational comparison of subarachnoid hemorrhage epidemiology in the WHO MONICA stroke study. Stroke. 2000;31:1054-61.). In this relative high mortality rate the effect of delayed cerebral ischaemia (DCI) and different extracerebral complications (Takotsubo cardiomyopathy, secondary infections, etc.) have key roles. (Claassen J, Vu A, Kreiter KT, et al. Effect of acute physiologic derangements on outcome after subarachnoid hemorrhage. Crit Care Med. 2004;32:832-8.). DCI occurs in nearly third of patients and its most common cause is cerebral vasospasm (at least 70% of cases). Vasospasm usually develops on day 3 after hemorrhage, it reaches a peak on day 7-8 and solves after the day 14.

(Dorsch NWC, King MT. A review of cerebral vasospasm in aneurysmal subarachnoid hemorrhage. Part 1: Incidence and effects. J Clin Neurosci. 1994;1:19-26.).

DCI has been shown to be a multifactorial process, in which cerebral vasospasm has a remarkable part, but anemia, cortical spreading depolarization, damage of cerebral autoregulation, and activation of the inflammatory-thrombotic cascade may also play an important role. . (Chamling B, Gross S, Stoffel-Wagner B, Schubert GA, Clusmann H, Coburn M, et al. Early diagnosis of delayed cerebral ischemia: possible relevance for inflammatory biomarkers in routine clinical practice? World Neurosurg (2017) 104:152-7. McBride DW, Blackburn SL, Peeyush KT, Matsumura K, Zhang JH. The Role of Thromboinflammation in Delayed Cerebral Ischemia after Subarachnoid Hemorrhage.Front Neurol. 2017;8:555.).

In this prospective study the investigators aim to investigate the role of the following three factors on the development of vasospasm and patient outcome: (1.) anemia; (2.) plasma fibrinolytic activity; (3.) vitamin D.

Review of related literature:

The role of anaemia in SAH: Depending on definition, anaemia develops in 40-50% of SAH patients, only 16% of patients have a hemoglobin level higher than 110g/l . According to follow-up studies anaemia appears on day 3-4 after hemorrhage (concurrently with vasospasm) and the reduction of hemoglobin concentration is 30 g/l on average. (Sampson TR, Dhar R, Diringer MN. Factors associated with the development of anemia after subarachnoid hemorrhage. Neurocrit Care. 2010;12:4-9.)

Clot lysis assay gives an opportunity to detect the plasma fibrinolytic potential. Studies from the recent years identified neutrophil extracellular trap (NET) components, releasing from activated neutrophil granulocytes and play an important role in the modulation of the fibrinolytic process. NETs are the part of the complex system of inherited immunity. A recent study has shown that parameters of the modified CLA correlate with the volume of hematoma and outcome of spontaneous intracranial hemorrhage. (Orbán-Kálmándi R, Árokszállási T, Fekete I, Fekete K, Héja M, Tóth J, Sarkady F, Csiba L, Bagoly Z. A Modified in vitro Clot Lysis Assay Predicts Outcomes in Non-traumatic Intracerebral Hemorrhage Stroke Patients-The IRONHEART Study. Front Neurol. 2021;12:613441.) No similar studies exist about SAH.

The role of vitamine D3 in SAH: In a previous pilot study vitamine D3 deficiency was identified as an independent risk factor of SAH outcome , furthermore vitamin D3 level was inversely related to the incidence and severity of vasospasm. (Kashefiolasl S, Leisegang MS, Helfinger V, Schürmann C, Pflüger-Müller B, Randriamboavonjy V, Vasconez AE, Carmeliet G, Badenhoop K, Hintereder G, Seifert V, Schröder K, Konczalla J, Brandes RP. Vitamin D-A New Perspective in Treatment of Cerebral Vasospasm. Neurosurgery. 2021;88:674-685.).

Perspectives of the planned study: Considering the currently available therapeutic range for patients with SAH, results of the present study may provide a basis for designing further randomized, prospective trials to investigate the effect of treating anemia, anticoagulation and vitamin D supplementation.

Subjects and methods

The investigators include patients admitted to the Neurosurgical Intensive Care Unit of the Clinical Center of the University of Debrecen with the diagnosis of SAH.

Inclusion criteria:

* acut SAH
* patients older than 18 years
* admission within 48 hours after symptom onset

Exclusion criteria:

* admission over 48 hours after symptom onset
* traumatic SAH
* Angioma
* A-V malformation
* Patient unable to consent and no relative available

Planned period of patient enrollment: June 1, 2022 - December 31, 2024 Planned number of patients: approx. 300 patients

Patients are treated according to local protocol based on international guidelines(Diringer MN, Bleck TP, Claude Hemphill J 3rd, Menon D, Shutter L, Vespa P, Bruder N, Connolly ES Jr, Citerio G, Gress D, Hänggi D, Hoh BL, Lanzino G, Le Roux P, Rabinstein A, Schmutzhard E, Stocchetti N, Suarez JI, Treggiari M, Tseng MY, Vergouwen MD, Wolf S, Zipfel G; Neurocritical Care Society. Critical care management of patients following aneurysmal subarachnoid hemorrhage: recommendations from the Neurocritical Care Society's Multidisciplinary Consensus Conference. Neurocrit Care. 2011;15:211-240.), and neurosurgeons and interventional radiologists are involved in therapeutic decisions.

Investigations and recorded data on admission:

* skull CT
* angiography
* severity classification: Fisher, Hunt-Hess, WFNS, GCS
* medical history, especially: hypertension, diabetes mellitus, cardiovascular diseases, kidney diseases (polycystic kidney? ), previous stroke
* laboratory investigations: blood count, blood glucose, kidney function, hemostasis + fibrinogen

Investigations associated with present study and their timing:

Hemoglobin level:

* day of admission
* day 3-4-7 and 14 after hemorrhage

mCLA:

* day of admission
* day 7 after hemorrhage

  25-hydroxy vitamin-D level:
* day of admission

Transcranial color- coded duplex sonography:

* daily basis

  30 day follow-up:
* mortality
* Glasgow Outcome Scale
* Karnofsky score
* Barthel score

  90 day follow-up:
* mortality
* Glasgow Outcome Scale
* Karnofsky score
* Barthel score

Transcranial color-coded duplex sonography :

Transcranial color-coded duplex (TCCD) sonography is performed by two experienced investigators (Béla Fülesdi, Péter Síró) using the 2 MHz sector transducer of the GE Venue Go (GE Healthcare 9900 Innovation Drive Wauwatosa, WI 53226 U.S.A.) ultrasound device. Regular TCCD measurements are registered in all patients between days 1 through 7. Based on previous suggestions, vasospasm is considered if mean blood flow velocity was higher than 120 cm/s and severe vasospasm is diagnosed if mean blood flow velocity exceeded 200 cm/s. If ultrasound signs of vasospasm are present in any of the cases, duplex sonographies are performed until day 21 on a daily basis.

Processing data

Correlation of all three parameters with SAV severity parameters, detected on admission: Hunt Hess score, Fischer score, WFNS score

Correlation of all three parameters with the development of vasospasm.

Definition of anemia based on hemoglobin level:

* in males: < 120 g / l
* in females: <110 g / l

  25-hydroxy vitamin-D level:
* definition of low level: <50 nmol/l

Statistical analysis:

To analyse continuous variables, in the first step a normality test is performed. The t-test is used to analyse samples with a normal distribution, while non-parametric tests are used to analyse samples with non-normal distribution. Bonferroni correction is performed for multiple comparisons. To examine categorical variables, the investigators use a χ2 test with "Yates' correction for continuity" if necessary.

ELIGIBILITY:
Inclusion Criteria:

* acut SAH
* patients older than 18 years
* admission within 48 hours after symptom onset

Exclusion Criteria:

* admission over 48 hours after symptom onset
* traumatic SAH
* Angioma
* A-V malformation
* Patient unable to consent and no relative available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study intends to include all patients over 18 years of age who were admitted to our clinic within 48 hours after the bleeding regardless of gender, neurological status or age.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin level | day of admission, day 3-4-7 and 14 after hemorrhage
  correlation with the development of vasospasm
mCLA | day of admission, day 7 after hemorrhage
  correlation with the development of vasospasm
25-hydroxy vitamin-D level | day of admission
  correlation with the development of vasospasm

SECONDARY OUTCOMES:
Hemoglobin level | day 14, 30 and 90 after hemorrhage
  correlation with outcome (GOS, Barthel Index, Karnofsky Index)
mCLA | day 14, 30 and 90 after hemorrhage
  correlation with outcome (GOS, Barthel Index, Karnofsky Index)
25-hydroxy vitamin-D level | day 14, 30 and 90 after hemorrhage
  correlation with outcome (GOS, Barthel Index, Karnofsky Index)

CONTACTS AND LOCATIONS:
Overall Officials: Csilla Molnár, MD Associate professor, Principal Investigator — Department of Anesthesiology and Intensive Care, University of Debrecen, Health and Medical Science Centre
Locations (1):
- Dr. Szántó Dorottya, Debrecen, Hajdú-Bihar, Hungary

REFERENCES:
- [Background] Etminan N, Chang HS, Hackenberg K, de Rooij NK, Vergouwen MDI, Rinkel GJE, Algra A. Worldwide Incidence of Aneurysmal Subarachnoid Hemorrhage According to Region, Time Period, Blood Pressure, and Smoking Prevalence in the Population: A Systematic Review and Meta-analysis. JAMA Neurol. 2019 May 1;76(5):588-597. doi: 10.1001/jamaneurol.2019.0006. PMID 30659573
- [Background] Epidemiology of aneurysmal subarachnoid hemorrhage in Australia and New Zealand: incidence and case fatality from the Australasian Cooperative Research on Subarachnoid Hemorrhage Study (ACROSS). Stroke. 2000 Aug;31(8):1843-50. doi: 10.1161/01.str.31.8.1843. PMID 10926945
- [Background] Ingall T, Asplund K, Mahonen M, Bonita R. A multinational comparison of subarachnoid hemorrhage epidemiology in the WHO MONICA stroke study. Stroke. 2000 May;31(5):1054-61. doi: 10.1161/01.str.31.5.1054. PMID 10797165
- [Background] Rowland MJ, Hadjipavlou G, Kelly M, Westbrook J, Pattinson KT. Delayed cerebral ischaemia after subarachnoid haemorrhage: looking beyond vasospasm. Br J Anaesth. 2012 Sep;109(3):315-29. doi: 10.1093/bja/aes264. PMID 22879655
- [Background] Claassen J, Vu A, Kreiter KT, Kowalski RG, Du EY, Ostapkovich N, Fitzsimmons BF, Connolly ES, Mayer SA. Effect of acute physiologic derangements on outcome after subarachnoid hemorrhage. Crit Care Med. 2004 Mar;32(3):832-8. doi: 10.1097/01.ccm.0000114830.48833.8a. PMID 15090970
- [Background] Dorsch NW, King MT. A review of cerebral vasospasm in aneurysmal subarachnoid haemorrhage Part I: Incidence and effects. J Clin Neurosci. 1994 Jan;1(1):19-26. doi: 10.1016/0967-5868(94)90005-1. PMID 18638721
- [Background] Chamling B, Gross S, Stoffel-Wagner B, Schubert GA, Clusmann H, Coburn M, Hollig A. Early Diagnosis of Delayed Cerebral Ischemia: Possible Relevance for Inflammatory Biomarkers in Routine Clinical Practice? World Neurosurg. 2017 Aug;104:152-157. doi: 10.1016/j.wneu.2017.05.021. Epub 2017 May 13. PMID 28512045
- [Background] McBride DW, Blackburn SL, Peeyush KT, Matsumura K, Zhang JH. The Role of Thromboinflammation in Delayed Cerebral Ischemia after Subarachnoid Hemorrhage. Front Neurol. 2017 Oct 23;8:555. doi: 10.3389/fneur.2017.00555. eCollection 2017. PMID 29109695
- [Background] Sampson TR, Dhar R, Diringer MN. Factors associated with the development of anemia after subarachnoid hemorrhage. Neurocrit Care. 2010 Feb;12(1):4-9. doi: 10.1007/s12028-009-9273-1. Epub 2009 Sep 24. PMID 19777386
- [Background] Orban-Kalmandi R, Arokszallasi T, Fekete I, Fekete K, Heja M, Toth J, Sarkady F, Csiba L, Bagoly Z. A Modified in vitro Clot Lysis Assay Predicts Outcomes in Non-traumatic Intracerebral Hemorrhage Stroke Patients-The IRONHEART Study. Front Neurol. 2021 Apr 20;12:613441. doi: 10.3389/fneur.2021.613441. eCollection 2021. PMID 33959087
- [Background] Kashefiolasl S, Leisegang MS, Helfinger V, Schurmann C, Pfluger-Muller B, Randriamboavonjy V, Vasconez AE, Carmeliet G, Badenhoop K, Hintereder G, Seifert V, Schroder K, Konczalla J, Brandes RP. Vitamin D-A New Perspective in Treatment of Cerebral Vasospasm. Neurosurgery. 2021 Feb 16;88(3):674-685. doi: 10.1093/neuros/nyaa484. PMID 33269399
- [Background] Diringer MN, Bleck TP, Claude Hemphill J 3rd, Menon D, Shutter L, Vespa P, Bruder N, Connolly ES Jr, Citerio G, Gress D, Hanggi D, Hoh BL, Lanzino G, Le Roux P, Rabinstein A, Schmutzhard E, Stocchetti N, Suarez JI, Treggiari M, Tseng MY, Vergouwen MD, Wolf S, Zipfel G; Neurocritical Care Society. Critical care management of patients following aneurysmal subarachnoid hemorrhage: recommendations from the Neurocritical Care Society's Multidisciplinary Consensus Conference. Neurocrit Care. 2011 Sep;15(2):211-40. doi: 10.1007/s12028-011-9605-9. PMID 21773873
- [Background] Maher M, Schweizer TA, Macdonald RL. Treatment of Spontaneous Subarachnoid Hemorrhage: Guidelines and Gaps. Stroke. 2020 Apr;51(4):1326-1332. doi: 10.1161/STROKEAHA.119.025997. Epub 2020 Jan 22. No abstract available. PMID 31964292